CLINICAL TRIAL: NCT04346342
Title: PRactice of VENTilation in COVID-19 Patients (PRoVENT-COVID) - an Observational Study of Invasively Ventilated Patients in the Netherlands
Brief Title: PRactice of VENTilation in COVID-19 Patients (PRoVENT-COVID)
Acronym: PRoVENT-COVID
Status: Completed | Type: Observational
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, Prof. Dr. Marcus J. Schultz, Prof., Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Other Study IDs: PRoVENT-COVID
Record Dates: First submitted 2020-04-09; First posted 2020-04-15 (Actual); Last update posted 2021-07-06 (Actual); Status verified 2021-07

CONDITIONS: COVID; Mechanical Ventilation; Acute Respiratory Failure
Keywords: COVID

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Mechanical ventilation: COVID patients receiving invasive mechanical ventilation

SUMMARY:
The purpose of this national, multicenter service review is to determine and compare ventilation management in COVID-19 patients in the Netherlands, and to determine whether certain ventilation settings have an independent association with duration of ventilation.

In every adult invasively ventilated COVID-19 patient from a participating ICU, granular ventilator settings and parameters will be collected from start of invasive ventilation for up to 72 hours. Follow up is until ICU and hospital discharge, and until day 90. The primary outcome includes main ventilator settings (including tidal volume, airway pressures, oxygen fraction and respiratory rate). Secondary endpoints are ventilator-free days and alive at day 28 (VFD-28); duration of mechanical ventilation; use of prone positioning and recruitment maneuvers; duration of ICU and hospital stay; incidence of kidney injury; and ICU, hospital, 28-day and 90-day mortality.

DETAILED DESCRIPTION:
Rationale:

The novel coronavirus disease (COVID-19) pandemic is rapidly expanding across the world, with over 60.000 new cases each day as of late March 2020. Healthcare workers are struggling to provide the best care for patients with proven or suspected COVID-19. Approaches for clinical care vary widely between and within countries and new insights are acquired rapidly. This includes the way invasive ventilation is applied.

Objective:

To determine and compare invasive ventilation settings and parameters in COVID-19 patients in the Netherlands, and to determine associations with clinical outcomes.

Hypotheses:

Invasive ventilation settings and parameters vary between intensive care units (ICUs) in hospitals in the Netherlands; certain ventilator settings have an independent association with duration of ventilation in COVID-19 patients.

Study design:

Multicenter, national, retrospective, observational study in COVID-19 patients with respiratory failure, requiring invasive ventilation in intensive care unit (ICU) in hospitals in the Netherlands.

Study population:

The data of at least 1,000 consecutively invasively ventilated COVID-19 patients admitted to intensive care units (ICUs) of hospitals in the Netherlands. This study will not be restricted to the 'formal' ICUs, as patients may also receive invasive ventilation in other locations within the hospital during the COVID-19 pandemic.

Methods:

In every patient, granular ventilator settings and parameters are collected from start of invasive ventilation for up to 72 hours. Patients will be followed up until ICU and hospital discharge, and until day 90.

Sample size calculation:

No formal sample size calculation is needed. We expect to capture at least 1,000 patients, but will continue collecting data of new patients for at least 8 weeks.

Study endpoints:

Main ventilator settings (including tidal volume, airway pressures, oxygen fraction and respiratory rate) (primary) and parameters (blood gas results); use of rescue therapies (including prone positioning); use of sedatives, vasopressors and inotropes; daily cumulative fluid balances; development of kidney injury; ventilator-free days and alive at day 28 (VFD-28), duration of ICU and hospital stay, and ICU, hospital and 90-day mortality.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness:

Retrospective collection of data regarding ventilation management and major clinical endpoints is without risk for the individual patient.

ELIGIBILITY:
Inclusion Criteria:

* COVID-19, confirmed with polymerase chain reaction (PCR) and/or presence of typical abnormalities on chest computer tomography (CT)
* Suspected COVID-19 infection, with no exclusion of diagnosis
* Having received invasive ventilation

Exclusion Criteria:

* Age <18 years
* Already included in the same study in another hospital
* Having had received invasive ventilation > 24 hours in a non-participating hospital

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Invasively ventilated patients with COVID-19.
Sampling Method: Non-Probability Sample
Enrollment: 1122 (Actual)
Dates: Start 2020-03-06 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2020-09-01 (Actual)

PRIMARY OUTCOMES:
Ventilation Mode | Day 1 to Day 3 from initiation of mechanical ventilation
Tidal volume set | Day 1 to Day 3 from initiation of mechanical ventilation
Expiratory tidal volume | Day 1 to Day 3 from initiation of mechanical ventilation
Positive end-expiratory pressure | Day 1 to Day 3 from initiation of mechanical ventilation
Maximum airway pressure or plateau pressure (P plateau) or peak pressure (P peak) (cm H2O); | Day 1 to Day 3 from initiation of mechanical ventilation
Level of pressure support above positive end-expiratory pressure (PEEP) | Day 1 to Day 3 from initiation of mechanical ventilation
Inspired fraction of oxygen | Day 1 to Day 3 from initiation of mechanical ventilation
Set and measured respiratory rate | Day 1 to Day 3 from initiation of mechanical ventilation
Inspiration to expiration ratio | Day 1 to Day 3 from initiation of mechanical ventilation

SECONDARY OUTCOMES:
Number of ventilation-free days and alive at day 28 | Until 28 days from initiation of mechanical ventilation
Duration of ventilation in survivors; | Until 28 days from initiation of mechanical ventilation
  time between start invasive ventilation and successful extubation in survivors
Use of prone positioning | Day 1 to Day 3 from initiation of mechanical ventilation
Use of recruitment maneuvers | Day 1 to Day 3 from initiation of mechanical ventilation
Incidence of acute kidney injury | Until 28 days from initiation of mechanical ventilation
Duration of ICU stay | Until 28 days from initiation of mechanical ventilation
  Time between admission and discharge ICU or death in ICU
Duration of hospital stay | Until 28 days from initiation of mechanical ventilation
  Time between admission and discharge from hospital or death in hospital
ICU mortality | Until 28 days from initiation of mechanical ventilation
  Any death during ICU stay
Hospital mortality | Until 28 days from initiation of mechanical ventilation
  Any death during hospital stay
28-day mortality | Until 28 days from initiation of mechanical ventilation
90-day mortality | Until 90 days from initiation of mechanical ventilation

CONTACTS AND LOCATIONS:
Overall Officials: Marcus Schultz, MD, PhD, Principal Investigator — Department of Intensive Care, Academic Medical Center, University of Amsterdam; Frederique Paulus, PhD, Study Chair — Department of Intensive Care, Academic Medical Center, University of Amsterdam; Ary Serpa Neto, MD, PhD, Study Chair — Department of Intensive Care, Academic Medical Center, University of Amsterdam; Anna Geke Algera, MD, Study Director — Department of Intensive Care, Academic Medical Center, University of Amsterdam; Anissa Tsonas, MD, Study Director — Department of Intensive Care, Academic Medical Center, University of Amsterdam; Michela Botta, MD, Study Director — Department of Intensive Care, Academic Medical Center, University of Amsterdam
Locations (22):
- Netherlands (22):
  - Flevoziekenhuis, Almere Stad
  - Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA), Amsterdam
  - Onze Lieve Vrouwe Gasthuis, Amsterdam
  - Gelre ziekenhuizen, Apeldoorn
  - Rijnstate Ziekenhuis, Arnhem
  - Amphia Ziekenhuis, Breda
  - Reinier de Graaf Gasthuis, Delft
  - Ziekenhuis Gelderse Vallei, Ede
  - Catharina Ziekenhuis, Eindhoven
  - Maxima Medical Center, Eindhoven
  - St Anna Ziekenhuis, Geldrop
  - Universitair Medisch Centrum Groningen, Groningen
  - Spaarne Gasthuis, Haarlem
  - Dijklander Ziekenhuis, Hoorn
  - Leeuwarden Medisch Centrum, Leeuwarden
  - Maastricht Universitair Medisch Centrum, Maastricht
  - St Antonius Ziekenhuis, Nieuwegein
  - Maasstad Hospital, Rotterdam
  - Zuyderland Medisch Centrum, Sittard
  - Haaglanden Medisch Centrum, The Hague
  - HagaZiekenhuis, The Hague
  - Isala Ziekenhuis, Zwolle

REFERENCES:
- [Derived] Ahuja S, de Grooth HJ, Paulus F, van der Ven FL, Serpa Neto A, Schultz MJ, Tuinman PR; PRoVENT-COVID Study Collaborative Group* 'PRactice of VENTilation in COVID-19'. Association between early cumulative fluid balance and successful liberation from invasive ventilation in COVID-19 ARDS patients - insights from the PRoVENT-COVID study: a national, multicenter, observational cohort analysis. Crit Care. 2022 Jun 1;26(1):157. doi: 10.1186/s13054-022-04023-y. PMID 35650616
- [Derived] Schuijt MTU, van Meenen DMP, Martin-Loeches I, Mazzinari G, Schultz MJ, Paulus F, Serpa Neto A. Association of Time-Varying Intensity of Ventilation With Mortality in Patients With COVID-19 ARDS: Secondary Analysis of the PRoVENT-COVID Study. Front Med (Lausanne). 2021 Nov 18;8:725265. doi: 10.3389/fmed.2021.725265. eCollection 2021. PMID 34869421
- [Derived] Bos LDJ, Sjoding M, Sinha P, Bhavani SV, Lyons PG, Bewley AF, Botta M, Tsonas AM, Serpa Neto A, Schultz MJ, Dickson RP, Paulus F; PRoVENT-COVID collaborative group. Longitudinal respiratory subphenotypes in patients with COVID-19-related acute respiratory distress syndrome: results from three observational cohorts. Lancet Respir Med. 2021 Dec;9(12):1377-1386. doi: 10.1016/S2213-2600(21)00365-9. Epub 2021 Oct 13. PMID 34653374
- [Derived] Schuijt MTU, Schultz MJ, Paulus F, Serpa Neto A; PRoVENT-COVID Collaborative Group. Association of intensity of ventilation with 28-day mortality in COVID-19 patients with acute respiratory failure: insights from the PRoVENT-COVID study. Crit Care. 2021 Aug 6;25(1):283. doi: 10.1186/s13054-021-03710-6. PMID 34362415
- [Derived] Valk CMA, Tsonas AM, Botta M, Bos LDJ, Pillay J, Serpa Neto A, Schultz MJ, Paulus F; Writing Committee for the PRoVENT-COVID * Collaborative Group. Association of early positive end-expiratory pressure settings with ventilator-free days in patients with coronavirus disease 2019 acute respiratory distress syndrome: A secondary analysis of the Practice of VENTilation in COVID-19 study. Eur J Anaesthesiol. 2021 Dec 1;38(12):1274-1283. doi: 10.1097/EJA.0000000000001565. PMID 34238782
- [Derived] Boers NS, Botta M, Tsonas AM, Algera AG, Pillay J, Dongelmans DA, Horn J, Vlaar APJ, Hollmann MW, Bos LDJ, Paulus F, Neto AS, Schultz MJ; PRoVENT-COVID investigatorsdagger. PRactice of VENTilation in Patients with Novel Coronavirus Disease (PRoVENT-COVID): rationale and protocol for a national multicenter observational study in The Netherlands. Ann Transl Med. 2020 Oct;8(19):1251. doi: 10.21037/atm-20-5107. PMID 33178783
- [Derived] Botta M, Tsonas AM, Pillay J, Boers LS, Algera AG, Bos LDJ, Dongelmans DA, Hollmann MW, Horn J, Vlaar APJ, Schultz MJ, Neto AS, Paulus F; PRoVENT-COVID Collaborative Group. Ventilation management and clinical outcomes in invasively ventilated patients with COVID-19 (PRoVENT-COVID): a national, multicentre, observational cohort study. Lancet Respir Med. 2021 Feb;9(2):139-148. doi: 10.1016/S2213-2600(20)30459-8. Epub 2020 Oct 23. PMID 33169671

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-06-01): https://cdn.clinicaltrials.gov/large-docs/42/NCT04346342/Prot_SAP_001.pdf